CLINICAL TRIAL: NCT00174655
Title: An Intergroup Phase III Trial to Evaluate the Activity of Docetaxel, Given Either Sequentially or in Combination With Doxorubicin, Followed by CMF, in Comparison to Doxorubicin Alone or in Combination With Cyclophosphamide, Followed by CMF, in the Adjuvant Treatment of Node-positive Breast Cancer Patients.
Brief Title: BIG 02/98 Docetaxel - Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP56976_PR_315; NCT00005659 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin

ARMS (4):
- A1 (Active Comparator)
  Interventions: Drug: doxorubicine + cyclophosphamide sequential
- A2 (Active Comparator)
  Interventions: Drug: doxorubicine + cyclophosphamide combined
- B (Experimental)
  Interventions: Drug: Doxorubicine + docetaxel sequential
- C (Experimental)
  Interventions: Drug: doxorubicine + docetaxel combined

INTERVENTIONS:
Drug: Doxorubicine + docetaxel sequential — doxorubicin 75 mg/m² i.v. day 1, q 21 days for 3 cycles, followed by docetaxel 100 mg/m² i.v., 1 hour infusion, day 1, q 21 days for 3 cycles, followed by CMF for 3 cycles
  Arms: B
Drug: doxorubicine + cyclophosphamide sequential — doxorubicin 75 mg/m² i.v. day 1 q 21 days for 4 cycles, followed by CMF (C: cyclophosphamide 100 mg/m² orally days 1-14, M: methotrexate: 40 mg/m² i.v. days 1 and 8, FU; 5-fluorouracil: 600 mg/m²) i.v. days 1 and 8, q 28 days for 3 cycles
  Arms: A1
Drug: doxorubicine + cyclophosphamide combined — doxorubicin 60 mg/m² i.v. + cyclophosphamide 600 mg/m² i.v., day 1, q 21 days for 4 cycles, followed by CMF for 3 cycles.
  Arms: A2
Drug: doxorubicine + docetaxel combined — doxorubicin 50 mg/m² i.v. + docetaxel 75 mg/m² i.v. 1 hour infusion (1 hour after doxorubicin), day 1, q 21 days for 4 cycles, followed by CMF for 3 cycles.
  Arms: C

SUMMARY:
Primary objectives:

* To compare Disease-Free Survival (DFS) of an adjuvant treatment with docetaxel given either sequentially or in combination with doxorubicin and followed by CMF to doxorubicin alone or in combination with cyclophosphamide and followed by CMF in operable breast cancer patients with positive axillary lymph nodes.

Secondary objectives:

* To compare DFS of an adjuvant treatment with doxorubicin followed by docetaxel followed by CMF to doxorubicin followed by CMF in operable breast cancer patients with positive axillary lymph nodes
* To compare DFS of an adjuvant treatment with docetaxel in combination with doxorubicin followed by CMF to doxorubicin in combination with cyclophosphamide followed by CMF in operable breast cancer patients with positive axillary lymph nodes
* To compare DFS of an adjuvant treatment with doxorubicin followed by docetaxel followed by CMF to doxorubicin in combination with docetaxel followed by CMF in operable breast cancer patients with positive axillary lymph nodes, (sequential mono-chemotherapy versus polychemotherapy).
* To compare overall survival of treatment arms.
* To compare toxicity of treatment arms.
* To evaluate pathologic and molecular markers for predicting efficacy.
* Socioeconomic data will be collected in order to be able to perform a socioeconomic analysis by country, when needed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven breast cancer. Interval between definitive surgery that includes axillary lymph node dissection and registration must be less than 60 days. A representative sample of the primary tumor (either blocks or slides) must be sent to the operational office, for central pathology reviews, after patients randomization.
* Definitive surgical treatment must be either mastectomy or breast conserving surgery, with axillary lymph node dissection (not sampling) for operable breast cancer (clinical T1-3, N0-1, M0). Margins of resected specimen from definitive surgery must be histologically free of invasive adenocarcinoma and ductal carcinoma in situ (DCIS). Lobular carcinoma in-situ does not count as a positive margin. Patients with histologically-documented infiltration of the skin (pT4) will not be eligible. Patients who have a breast conserving procedure with a positive margin may become eligible if they subsequently undergo adequate resection or mastectomy with clear margins.
* Histologic examination of the tumor: invasive adenocarcinoma with at least one axillary lymph node (pN1) showing evidence of tumor among a minimum of eight resected lymph nodes. All nodes must be examined by the pathologist. The determination of ER (estrogen receptor) and PgR (progesterone receptor) is mandatory and results must be known by the end of chemotherapy in order to decide whether hormonal therapy is indicated (Biochemical or immunohistochemical methods required ; ER and/or PgR positivity should be in accordance with the policy in use at each participating center. Each center will specify its own policy).
* Age > or = 18 years and age < or = 70 years. The upper age limit is not meant to be exclusionary but rather is based on the lack of safety data for women > 70 years of age.
* Karnofsky Performance status index > or = 70 %.
* Normal cardiac function must be confirmed by LVEF (MUGA scan or echocardiography). The result must be above the lower limit of normal for the institution.
* Laboratory requirements: (within 14 days prior to registration)

  * Hematology

    * Neutrophils > or = 2.0 x 109/L
    * Platelets > or =100 x 109/L
    * Hemoglobin > or = 10 g/dL
  * Hepatic function

    * Total bilirubin < or = 1 UNL
    * ASAT (SGOT) and ALAT (SGPT) < or = 1.5 UNL
    * Alkaline phosphatase < or = 2.5 UNL
  * Renal function

    * Creatinine < or = 150 µmol/L (1.5 mg/dL)
    * If creatinine is borderline, the calculated creatinine clearance should be > or = 60 mL/min (Cockcroft formula).
* Complete staging work-up within 3 months prior to registration. All patients will have bilateral mammography, chest X-ray (PA and lateral) and/or CT-scan, abdominal ultrasound and/or CT scan, bone scan (in case of positive bone scan suspicious for metastases, bone X-ray (or bone CT-scan for spine) on hot spots is mandatory to rule out the possibility of metastatic hot spots). Other tests may be performed as clinically indicated.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at a participating center which could be a Principal or a co-investigator's site. In case patient moves during the follow-up, every effort should be done to follow the patient in a participating center.
* Negative pregnancy test (urine or serum) within 7 days prior to registration for all women of childbearing potential. Patients of childbearing potential must implement adequate non-hormonal measures to avoid pregnancy during study treatment(chemotherapy, radiotherapy and hormonal therapy).

Exclusion Criteria:

* Prior systemic anticancer therapy for breast cancer (chemo-immuno-hormonotherapy).
* Prior radiation therapy for breast cancer.
* Pregnant, or lactating patients.
* Any locally advanced (clinical or pathological T4 and/or N2-known N3) or metastatic(M1) breast cancer.Patients with inoperable residual axillary nodal disease or with supraclavicular nodes.
* Pre-existing motor or sensory neurotoxicity of a severity ³ grade 2 by NCI criteria.
* Other serious illness or medical condition:

  * congestive heart failure or unstable angina pectoris, previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or high-risk uncontrolled arrhythmias
  * history of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
  * active uncontrolled infection
  * active peptic ulcer, unstable diabetes mellitus
* Past or current history of other neoplasms except for:

  * curatively treated basal cell skin cancer
  * adequately treated in situ carcinoma of the cervix
* In regard to past or current history of other breast carcinoma, criteria of exclusion are:

  * past history of ipsilateral or past or current history of contralateral invasive breast carcinoma
  * past or current history of contralateral ductal in situ breast carcinoma

A past or current history of ipsilateral ductal in situ or lobular in situ (ipsilateral or contralateral) breast carcinoma is not a criterion of exclusion.

* Chronic treatment with corticosteroids unless initiated > 6 months prior to study entry and at low dose (< or = 20 mg methylprednisolone or equivalent).
* Concurrent treatment with hormonal replacement therapy. Prior treatment should be stopped before study entry.
* Definite contraindications for the use of corticosteroids.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
* Concurrent treatment with any other anti-cancer therapy.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2887 (Actual)
Dates: Start 1998-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
DFS of docetaxel arms versus non toxanes arm (DFS: interval from the date of randomization to the date of local, regional or metastatic relapse or the date of second primary cancer or death for any cause whichever occurs first. | 810 events or median 5 year follow-up whichever occurs first

SECONDARY OUTCOMES:
DFS sequential/combined arms | 810 events or median 5 year follow-up whichever occurs first
Safety NCI common toxicity criteria | from baseline to study end

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Aussel, Study Director — Sanofi
Locations (21):
- Sanofi-Aventis, Macquarie Park, Australia
- Sanofi-Aventis, Vienna, Austria
- Sanofi-Aventis, Diegem, Belgium
- Sanofi-Aventis, São Paulo, Brazil
- Sanofi-Aventis, Providencia Santiago, Chile
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Hørsholm, Denmark
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Budapest, Hungary
- Sanofi-Aventis, Dublin, Ireland
- Sanofi-Aventis, Netanya, Israel
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, Auckland, New Zealand
- Sanofi-Aventis, Porto Salvo, Portugal
- Sanofi-Aventis, Bratislava, Slovakia
- Sanofi-Aventis, Ljubljana, Slovenia
- Sanofi-Aventis, Gauteng, South Africa
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Bromma, Sweden
- Sanofi-Aventis, Geneva, Switzerland
- Sanofi-Aventis, Guildford Surrey, United Kingdom

REFERENCES:
- [Derived] Desmedt C, Fornili M, Clatot F, Demicheli R, De Bortoli D, Di Leo A, Viale G, de Azambuja E, Crown J, Francis PA, Sotiriou C, Piccart M, Biganzoli E. Differential Benefit of Adjuvant Docetaxel-Based Chemotherapy in Patients With Early Breast Cancer According to Baseline Body Mass Index. J Clin Oncol. 2020 Sep 1;38(25):2883-2891. doi: 10.1200/JCO.19.01771. Epub 2020 Jul 2. PMID 32614702
- [Derived] Fernandez-Cuesta L, Oakman C, Falagan-Lotsch P, Smoth KS, Quinaux E, Buyse M, Dolci MS, Azambuja ED, Hainaut P, Dell'orto P, Larsimont D, Francis PA, Crown J, Piccart-Gebhart M, Viale G, Leo AD, Olivier M. Prognostic and predictive value of TP53 mutations in node-positive breast cancer patients treated with anthracycline- or anthracycline/taxane-based adjuvant therapy: results from the BIG 02-98 phase III trial. Breast Cancer Res. 2012 May 2;14(3):R70. doi: 10.1186/bcr3179. PMID 22551440